CLINICAL TRIAL: NCT06696521
Title: A Prospective Analysis of Medication Adherence Comparing Televideo and Telephonic Modes of Longitudinal Monitoring and Utilization of a Standardized Educational Protocol
Brief Title: An Analysis of Medication Adherence Using Televideo and Telephonic Monitoring and Utilization of an Education Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Principal Investigator, Elizabeth Prechtel Dunphy, DNP, RN, ANP-BC, AOCN, DNP, CRNP, Abramson Cancer Center at Penn Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UPCC24220
Record Dates: First submitted 2024-09-18; First posted 2024-11-20 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-11

CONDITIONS: Adherence, Medication; Cancer
MeSH Terms: conditions — Medication Adherence; Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients randomized to telephonic or televideo participation once enrolled in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Telephonic and telemedicine evaluation (Other): Patients will be randomized to telephonic or telemedicine evaluation during participation in the study
  Interventions: Behavioral: Intervention A- Telephone; Behavioral: Intervention B- Televideo

INTERVENTIONS:
Behavioral: Intervention A- Telephone — For intervention A: Once a patient is randomized to telephone (Intervention A), s/he will be scheduled for the series of follow up encounters via the assigned modality. The first interaction will occur within 72 hours of the patient receiving their prescribed OCA(s) at which time the standardized educational information regarding the agent(s), dosing of the medication and potential medication side effects will be reviewed with the patient and/or caregiver. The second through eighth encounters will take place every 2 weeks thereafter through the study timeframe up to four months to assess for adherence and toxicity. At each visit, an adherence assessment including pill count, and Oral Chemotherapy Adherence Scale (OCAS), fill history will be obtained prior to each interaction to verify medication possession ratio (MPR) and proportion of days covered (PDC). Each patient in the study will participate for a duration of up to 4 months.
Behavioral: Intervention B- Televideo — For intervention B: Once a patient is randomized to televideo (Intervention B), s/he will be scheduled for the series of follow up encounters via the assigned modality. The first interaction will occur within 72 hours of the patient receiving their prescribed OCA(s) at which time the standardized educational information regarding the agent(s), dosing of the medication and potential medication side effects will be reviewed with the patient and/or caregiver. The second through eighth encounters will take place every 2 weeks thereafter through the study timeframe up to four months to assess for adherence and toxicity. At each visit, an adherence assessment including pill count, and Oral Chemotherapy Adherence Scale (OCAS), fill history will be obtained prior to each interaction to verify medication possession ratio (MPR) and proportion of days covered (PDC). Each patient in the study will participate for a duration of up to 4 months.

SUMMARY:
The objective of this study is to evaluate adherence to oral oncologic medication regimens utilizing a standardized education tool to explain the dosing, side effects and purpose of oral chemotherapy via televideo or telephonic interactions. Researchers aim to evaluate whether the modality of education and monitoring impact adherence.

DETAILED DESCRIPTION:
The study will consist of eight total interactions. We will allow for a 72 hour window for each encounter to allow for patient flexibility and scheduling. The first encounter will include medication education using the standardized tool. The remaining seven interactions will include toxicity and adherence assessment through patient interviews, the OCAS, pill counts, and pharmacy fill data. All interactions will be completed via telephonic outreach or televideo platform by either CRNP, PA-C or PharmD. The patient will be approached when an OCA is prescribed to be given a copy of the OncoLink® patient education material and consent form for review. Patients will be randomized 1:1 to either televideo or telephonic interactions using a block size of 4. All study staff will be blinded to block size. Once a patient is randomized, s/he will be scheduled for the series of follow up encounters via the assigned modality. The first telemedicine interaction will occur within 72 hours of the patient receiving their prescribed OCA(s) at which time the standardized educational information regarding the agent(s), dosing of the medication and potential medication side effects will be reviewed with the patient and/or caregiver. The second encounter will occur approximately 2 weeks after the patient starts the medication to assess for adherence and toxicity. The third through eighth encounters will take place every 2 weeks thereafter through the study timeframe up to four months. At each visit, an adherence assessment including pill count, and Oral Chemotherapy Adherence Scale (OCAS) (Bagcivan and Akbayrak 2015) will be completed per standard of care in addition to patient interview to assess adherence and toxicity. Fill history will be obtained prior to each interaction to verify medication possession ratio and proportion of days covered.

Each patient in the study will participate for a duration of up to 4 months. All of the research will take place at the Abramson Cancer Center at Penn Presbyterian Medical Center.

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of cancer
2. Receives cancer care at Abramson Cancer Center at Penn Presbyterian Medical Center
3. Physically and cognitively able to provide informed consent
4. Is 18 years or older
5. Is starting an oral cancer agent
6. Has access to the UPENN televideo platform
7. Lives in Pennsylvania

Exclusion Criteria:

1. Does not desire to participate in the study
2. Cannot consent for himself/herself
3. Does not have access to the UPENN televideo platform
4. Does not live in Pennsylvania
5. Chemoradiation patients

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Will modality of outreach impact adherence based on medication possession ratio (MPR) or proportion of days covered (PDC)? | Through study completion, approximately 4 months
  The MPR and PDC will be calculated along with pill count and OCAS with each interaction through study completion and then evaluated for the individual patient and as an aggregate for all participants.
Will modality of outreach impact adherence based on medication pill counts? | Through study completion, approximately 4 months
  This will be measured with patient providing pill count at time of each interaction. MPR and PDC will also be calculated with each interaction to determine patient's compliance evaluating medication fill/refill information.
Will modality of outreach impact adherence based on Oral Chemotherapy Adherence Scale (OCAS)? | Through study completion, approximately 4 months
  The OCAS will be completed with each interaction and scored using the grading criteria of the scale authors. The OCAS scale contains 19 questions that are graded from 1-5 based on answer for a total score. A score of 84 and higher is classified as good adherence and a score of 83 and lower is classified as bad adherence. The highest score is 95 and the lowest score is 19. This calculation will be made with each interaction through the study completion. The scores will be analyzed for each patient and as an aggregate and compared between the groups

CONTACTS AND LOCATIONS:
Locations (1):
- Abramson Cancer Center at PPMC, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vrijens B, De Geest S, Hughes DA, Przemyslaw K, Demonceau J, Ruppar T, Dobbels F, Fargher E, Morrison V, Lewek P, Matyjaszczyk M, Mshelia C, Clyne W, Aronson JK, Urquhart J; ABC Project Team. A new taxonomy for describing and defining adherence to medications. Br J Clin Pharmacol. 2012 May;73(5):691-705. doi: 10.1111/j.1365-2125.2012.04167.x. PMID 22486599
- [Background] Voils CI, Venne VL, Weidenbacher H, Sperber N, Datta S. Comparison of Telephone and Televideo Modes for Delivery of Genetic Counseling: a Randomized Trial. J Genet Couns. 2018 Apr;27(2):339-348. doi: 10.1007/s10897-017-0189-1. Epub 2017 Dec 15. PMID 29243007
- [Background] Tipton JM. Overview of the challenges related to oral agents for cancer and their impact on adherence. Clin J Oncol Nurs. 2015 Jun;19(3 Suppl):37-40. doi: 10.1188/15.S1.CJON.37-40. PMID 26030391
- [Background] Spoelstra SL, Rittenberg CN. Assessment and measurement of medication adherence: oral agents for cancer. Clin J Oncol Nurs. 2015 Jun;19(3 Suppl):47-52. doi: 10.1188/15.S1.CJON.47-52. PMID 26030393
- [Background] Spoelstra SL, Given CW. Assessment and measurement of adherence to oral antineoplastic agents. Semin Oncol Nurs. 2011 May;27(2):116-32. doi: 10.1016/j.soncn.2011.02.004. PMID 21514481
- [Background] Sirintrapun SJ, Lopez AM. Telemedicine in Cancer Care. Am Soc Clin Oncol Educ Book. 2018 May 23;38:540-545. doi: 10.1200/EDBK_200141. PMID 30231354
- [Background] Burhenn PS, Smudde J. Using tools and technology to promote education and adherence to oral agents for cancer. Clin J Oncol Nurs. 2015 Jun;19(3 Suppl):53-9. doi: 10.1188/15.S1.CJON.53-59. PMID 26030395
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] McCabe CC, Barbee MS, Watson ML, Billmeyer A, Lee CE, Rupji M, Chen Z, Haumschild R, El-Rayes B. Comparison of rates of adherence to oral chemotherapy medications filled through an internal health-system specialty pharmacy vs external specialty pharmacies. Am J Health Syst Pharm. 2020 Jul 7;77(14):1118-1127. doi: 10.1093/ajhp/zxaa135. PMID 32537656
- [Background] Jacobs JM, Ream ME, Pensak N, Nisotel LE, Fishbein JN, MacDonald JJ, Buzaglo J, Lennes IT, Safren SA, Pirl WF, Temel JS, Greer JA. Patient Experiences With Oral Chemotherapy: Adherence, Symptoms, and Quality of Life. J Natl Compr Canc Netw. 2019 Mar 1;17(3):221-228. doi: 10.6004/jnccn.2018.7098. PMID 30865917
- [Background] Bertsch NS, Bindler RJ, Wilson PL, Kim AP, Ward B. Medication Therapy Management for Patients Receiving Oral Chemotherapy Agents at a Community Oncology Center: A Pilot Study. Hosp Pharm. 2016 Oct;51(9):721-729. doi: 10.1310/hpj5109-721. PMID 27803501
- [Background] Bagcivan G, Akbayrak N. Development and Psychometric Testing of the Turkish-Version Oral Chemotherapy Adherence Scale. J Nurs Res. 2015 Dec;23(4):243-51. doi: 10.1097/JNR.0000000000000101. PMID 26562455